CLINICAL TRIAL: NCT02640690
Title: Trauma-sensitive Yoga for Female Veterans With PTSD Who Experienced Military Sexual Trauma
Acronym: PSLII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRI 15-151
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Stress Disorders, Post-traumatic
Keywords: Stress Disorders, Post-traumatic; Yoga; Cognitive Therapy; Chronic Pain; Veterans; cytokines; acoustic startle reflex; women; heart rate variability; sexual trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain; Sexual Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma Center Trauma-Sensitive Yoga (TCTSY) (Experimental): 10-weekly 1-hour TCTSY Sessions
  Interventions: Behavioral: Trauma Center Trauma Sensitive Yoga Intervention (TCTSY)
- Cognitive Processing Therapy (CPT) (Active Comparator): 12-weekly 1.5 hour CPT Sessions
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Trauma Center Trauma Sensitive Yoga Intervention (TCTSY) — (10) 1-hour sessions of trauma sensitive yoga
  Arms: Trauma Center Trauma-Sensitive Yoga (TCTSY)
Behavioral: Cognitive Processing Therapy — (12) 1.5 hour sessions of cognitive processing therapy
  Other Names: Cognitive Processing Therapy-Cognitive
  Arms: Cognitive Processing Therapy (CPT)

SUMMARY:
In this study, we are evaluating the effectiveness of a yoga intervention to treat posttraumatic stress disorder (PTSD), its associated symptoms of chronic pain and insomnia, and biological and physiological responses to trauma and PTSD in women Veterans who experienced military sexual trauma (MST). If effective, this yoga intervention could reduce PTSD symptoms and chronic pain, improve sleep quality, and decrease the body's automatic "fight or flight" stress response and the damage this stress response causes in the body, including heart disease and diabetes. This intervention could improve these women Veterans' quality of life and social functioning, for example, going to work and having satisfying relationships with family and friends. This study may support an innovative, complementary and alternative PTSD treatment for women Veterans who experienced MST. This new, evidence-based PTSD treatment could supplement current PTSD treatments. Clinical guidelines for this yoga intervention could be implemented nationally in the VA health care system.

DETAILED DESCRIPTION:
Objectives: The overall goal of this project is to maximize the health, social functioning, and quality of life of women Veterans with posttraumatic stress disorder (PTSD) who have experienced military sexual trauma (MST). The specific aims of this randomized controlled trial (RCT) are to evaluate the effectiveness of a trauma-sensitive yoga intervention designed specifically for women who experienced sexual trauma as compared to a gold-standard PTSD treatment, Cognitive Processing Therapy, to 1) treat PTSD and its co-morbid symptoms of chronic pain and insomnia, 2) improve social functioning and quality of life, and 3) reduce the biological and psychophysiologic responses associated with PTSD in women Veterans who experienced MST.

Research Plan: This five year RCT is the next step following the NRI Pilot Study (NRI 12-417) in which the investigators demonstrated the feasibility of recruitment, retention, randomization, intervention implementation, and data collection, including biological and psychophysiological data. Women Veterans seeking treatment for PTSD were recruited from a primary site (southeast US) and second site (northwest US) and were randomized to Trauma Center Trauma-Sensitive Yoga (TCTSY) (10 weekly sessions) or Cognitive Processing Therapy (CPT) (12 weekly sessions); both intervention protocols are data-driven. The target enrollment sample size is 210, with a target final sample of 100 or more. The investigators are conservatively allowing for 50%-60% retention, based on pilot study results.

Methods: Data Collection: Data are collected at four points, baseline through 3-months post-intervention. Outcome measures include self-report, clinical assessments and biologic and psychophysiologic markers. Specific outcomes include PTSD symptom severity, chronic pain, insomnia, social functioning, quality of life, cytokines (IL-6, IL-10), C-reactive protein, heart rate variability, and dark-enhanced startle. Data Analysis: Comparisons between the groups at baseline will be run using t-tests, Mann Whitney non-parametric tests, and chi-square tests as appropriate. Multilevel mixed models (MLM) will be used to analyze the differences between the groups over time. MLM adjusts for attrition (missing data) over time and applies appropriate correlation structure between the time points.

Clinical Relevance: Women Veterans experience MST and PTSD at alarming rates; consistently reported prevalence rates for both among VHA patient samples are 20% or more. MST and PTSD put this population at risk for significant physical and mental health symptoms, including chronic pain, suicide, and negative health behaviors. This RCT may provide sufficient evidence to support an innovative, complementary and alternative PTSD treatment for women Veterans who experienced MST. The positive effects of reducing distressing symptoms and PTSD-related psychophysiological stress would likely improve social functioning and quality of life and minimize the significant medical consequences of PTSD in this population. This new, evidence-based PTSD treatment could supplement existing evidence-based PTSD treatment modalities. Clinical guidelines for this innovative intervention based on evidence from this clinical trial could be disseminated to and implemented in VA Medical Centers nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Women Veterans who experienced MST
* Diagnosed with PTSD related to MST
* Insomnia
* Willing to participate in either TCTSY or CPT study intervention

Exclusion Criteria:

* Schizophrenia with significant psychotic symptoms
* Current, active suicidal intent or plan
* Current substance abuse or dependence
* Certain medical conditions that can contribute significantly to psychiatric symptoms, including:

  * poorly controlled hypo/hyperthyroidism
  * kidney or liver failure
* Dementia
* Moderate or severe traumatic brain injury (TBI) or other cognitive impairment sufficient to interfere with ability to give informed consent
* Pain due to acute injury (<3 months), post-surgical pain (<3 months) or pain due to malignancy; pain related to injury and surgery are excluded to reduce risk of exacerbating underlying injury
* Receiving mental health treatment outside of the VA
* Ongoing participation in mental health treatment at odds with study intervention (For Example: yoga, trauma-focused treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A Kelly, PhD MSN BA, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaccari B, Loftis JM, Haywood T, Hubbard K, Clark J, Kelly UA. Synchronous Telehealth Yoga and Cognitive Processing Group Therapies for Women Veterans with Posttraumatic Stress Disorder: A Multisite Randomized Controlled Trial Adapted for COVID-19. Telemed J E Health. 2022 Mar 29:10.1089/tmj.2021.0612. doi: 10.1089/tmj.2021.0612. Online ahead of print. PMID 35357957
- [Background] Kelly U, Haywood T, Segell E, Higgins M. Trauma-Sensitive Yoga for Post-Traumatic Stress Disorder in Women Veterans who Experienced Military Sexual Trauma: Interim Results from a Randomized Controlled Trial. J Altern Complement Med. 2021 Mar;27(S1):S45-S59. doi: 10.1089/acm.2020.0417. PMID 33788599
- [Result] Zaccari B, Higgins M, Haywood TN, Patel M, Emerson D, Hubbard K, Loftis JM, Kelly UA. Yoga vs Cognitive Processing Therapy for Military Sexual Trauma-Related Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2344862. doi: 10.1001/jamanetworkopen.2023.44862. PMID 38064219
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 2016-2020 at two large Veterans Affairs (VA) Medical Centers in the US
Pre-assignment Details: 200 women consented. Additional assessments were conducted to confirm study eligibility. Women were considered protocol enrolled after study eligibility was confirmed. Of the 200, 35 did not meet inclusion criteria, 17 declined to participate prior to randomization, and 16 were lost to follow up, resulting in 132 women who were protocol enrolled and randomized; of those, one participant was administratively withdrawn (was enrolled in error). Thus, the final protocol enrollment was n=131.
Period: Overall Study
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Started | 72 | 59
Completed | 47 | 27
Not Completed | 25 | 32
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 16 | 20
Not completed — Partial completion (insufficient sessions) | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT) | Total
Number analyzed (Participants) | 72 | 59 | 131
Age, Categorical [Count of Participants; unit: Participants] — Self-reported age confirmed via medical records.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 67 | 57 | 124
    >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Full Range); unit: years] | 48.19 [26 to 70] | 48.27 [22 to 71] | 48.23 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported female sex at birth.
  Participants
    Female | 72 | 59 | 131
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 72 | 55 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 44 | 95
  White | 14 | 11 | 25
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 59 | 131
Clinician Assessed PTSD Scale-5 (CAPS-5) [Mean (Standard Deviation); unit: score on a scale] — CAPS-5 is a 30-item structured interview that can be used to assess PTSD symptom severity and presence or absence of criteria for PTSD diagnosis. Score with a possible range of 0-80. Higher scores mean worse outcome. Population: The CAPS-5 for two participants were incompletely scored by interviewer, therefore data are not usable.
  score on a scale
    number analyzed (Participants) | 71 | 58 | 129
    (all) | 36.73 (8.79) | 35.52 (7.49) | 36.19 (8.22)
PTSD Symptom Checklist (PCL-5) [Mean (Standard Deviation); unit: score on a scale] — PCL-5 is a 20-item measure of PTSD symptoms frequency. Total severity score ranging from 0-80, with higher scores representing greater symptom severity. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  score on a scale
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 49.62 (12.19) | 48.69 (13.62) | 49.20 (12.82)
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: score on a scale] — BDI-II is a 21-item self-report rating scale measuring the severity of depression symptoms. Score with a possible range of 0-63 with higher scores indicating worse outcomes. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Some participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 69 | 57 | 126
    (all) | 28.04 (9.83) | 28.98 (11.79) | 28.47 (10.72)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: score on a scale] — PSQI is a self-report scale consisting of 19 items that produces a global sleep quality score. Possible score ranges from 0-21 with higher score indicating worse outcome. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Four participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 69 | 57 | 126
    (all) | 14.07 (3.25) | 14.53 (3.08) | 14.28 (3.17)
Difficulties in Emotion Regulation Scale (DERS) [Mean (Standard Deviation); unit: score on a scale] — DERS is a brief 36-item, self-report questionnaire designed to assess multiple aspects of emotional dysregulation. Possible score ranges from 36-180 with higher scores indicating worse outcomes. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Three participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 71 | 56 | 127
    (all) | 92.10 (25.98) | 96.46 (23.58) | 94.03 (24.95)
BPI Pain Severity [Mean (Standard Deviation); unit: score on a scale] — The Brief Pain Inventory (BPI) Severity subscale contains three questions. Pain severity is measured according to the worst pain experienced in the last three days, average pain in the last three days, and current pain; with each rated on an ordinal scale from "0" = "no pain" to "10" = "pain as bad as you can imagine." The pain severity score is the mean of the three pain severity item scores, with a potential range of 0-10. Higher scores indicated worse outcomes. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Several participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 63 | 53 | 116
    (all) | 5.06 (2.00) | 5.28 (2.17) | 5.16 (2.07)
BPI Pain Interference [Mean (Standard Deviation); unit: score on a scale] — The Brief Pain Inventory (BPI) contains seven questions regarding pain interference that are rated on an ordinal numerical scale with anchors of 0 (no pain/interference) to 10 (maximum pain/interference). Pain interference assesses how that pain has affected general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. The pain interference score is the mean of the seven pain interference item scores, with a potential range of 0-10; higher scores indicate worse outcomes. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Several participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 63 | 53 | 116
    (all) | 4.90 (2.68) | 5.47 (2.49) | 5.16 (2.60)
DSM-5 Level 2-Somatic Symptom- adaptation of PHQ-15 (Patient Health Questionnaire Physical Symptoms) [Mean (Standard Deviation); unit: score on a scale] — This assesses the domain of somatic symptoms. The measure evaluates how often an individual has been bothered by a list of symptoms during the past 7 days. Possible scores range from 0-30 with higher scores indicating worse outcomes. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  score on a scale
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 13.22 (4.78) | 14.69 (4.39) | 13.89 (4.65)
PROMIS v2.0 Ability to Participate in Social Roles and Activities - Short Form 4a T-score [Mean (Standard Deviation); unit: T-score] — PROMIS v2.0 - Ability to Participate in Social Roles and Activities -Short Form 4a assesses the perceived ability to perform usual social roles and activities. Four items are worded negatively and are scored on a 5-point scale (5=never to 1= always). Responses are reverse-coded so that higher scores represent fewer limitations (better abilities). PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. A T-score higher than 50 indicates higher perceived ability to participate than the population mean. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  T-score
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 40.63 (7.25) | 41.00 (6.41) | 40.80 (6.86)
PROMIS v2.0 - Emotional Support -Short Form 4a T-Score [Mean (Standard Deviation); unit: T-score] — The PROMIS v2.0 - Emotional Support Short Form 4a assesses perceived feelings of being cared for, valued, and having confidant relationships using 4 items using a 5-point scale (1=never to 5=always). Per PROMIS scoring instructions, population-normed T-scores are used for analysis. Scores higher than 50 indicate more emotional support than the population mean. PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. A T-score higher than 50 indicates higher perceived emotional support than the population mean. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  T-score
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 46.78 (9.44) | 45.37 (10.70) | 46.14 (10.02)
PROMIS V2.0 Satisfaction with Social Roles and Activities - Short Form 4a T-score [Mean (Standard Deviation); unit: T-score] — The PROMIS V2.0 Satisfaction with Social Roles and Activities - Short Form 4a assesses satisfaction with performing social roles and activities using 4 items scored on a 5-point scale (1=not at all to 5=very much). PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. A T-score higher than 50 indicates higher satisfaction with social roles and activities than the population mean. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  T-score
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 39.92 (6.55) | 40.38 (7.72) | 40.13 (7.09)
PROMIS v2.0 - Social Isolation - Short Form 4a T-score [Mean (Standard Deviation); unit: T-score] — The PROMIS v2.0 - Social Isolation - Short Form 4a assesses perceptions of being avoided, excluded, detached, disconnected from or unknown by others, using 4 items scored on a five-point scale (1=never to 5=always). PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. A T-score higher than 50 indicates higher perceived social isolation than the population mean. Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study.
  T-score
    number analyzed (Participants) | 71 | 59 | 130
    (all) | 60.29 (8.14) | 59.17 (8.18) | 59.78 (8.14)
Health-related Quality of Life: Veterans Rand 12 (VR12) Mental Health [Mean (Standard Deviation); unit: score on a scale] — The VR-12 is a 12-item self-rating scale that assess health-related quality of life in veterans Results are expressed in terms of two meta-scores: the Mental Component Summary and the Physical Component Summary. The Mental Component Score (MCS) measures mental aspects of quality of life and ranges from 0 (extremely poor mental health) to 100 (extremely good mental health). The MCS is veteran population-normed with a mean score of 50 and a standard deviation of 10. Scores greater than 50 represent above average health status (better outcomes). Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Two participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 70 | 58 | 128
    (all) | 32.58 (11.32) | 30.69 (10.34) | 31.72 (10.88)
Health-related Quality of Life: Veterans Rand 12 (VR12) Physical Health [Mean (Standard Deviation); unit: score on a scale] — The VR-12 is a 12-item self-rating scale that assess health-related quality of life in veterans. Results are expressed in terms of two meta-scores: the Physical Component Summary and the Mental Component Summary. The Physical Component Score (PCS) measures physical aspects of quality of life and ranges from 0 (extremely poor physical health) to 100 (extremely good physical health), thus has a possible range of 0-100. The VR-12 is veteran population-normed with a mean score of 50 and a standard deviation of 10. Scores greater than 50 represent above average health status (better outcomes). Population: One TCTSY participant did not complete self-report measures at baseline, then withdrew from study. Several participants missed individual items in this measure, making their data unusable.
  score on a scale
    number analyzed (Participants) | 70 | 58 | 128
    (all) | 38.24 (11.82) | 37.66 (11.87) | 37.98 (11.80)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: LN(mg/L)] — Population: Some participants did not have blood samples drawn, resulting in missing data.
  LN(mg/L)
    number analyzed (Participants) | 55 | 38 | 93
    (all) | 0.73 (1.38) | 0.99 (1.28) | 0.83 (1.34)
Interleukin-6 (IL-6) Pro-inflammatory Cytokine [Mean (Standard Deviation); unit: LN(pg/mL)] — Population: Some participants did not have blood drawn, resulting in missing data.
  LN(pg/mL)
    number analyzed (Participants) | 55 | 38 | 93
    (all) | 1.05 (1.64) | 1.01 (1.56) | 1.03 (1.60)
Interleukin-10 (IL-10) Anti-inflammatory Cytokine [Mean (Standard Deviation); unit: LN(pg/mL)] — Population: Some participants did not have blood drawn, resulting in missing data.
  LN(pg/mL)
    number analyzed (Participants) | 55 | 38 | 93
    (all) | 2.59 (1.60) | 2.76 (1.76) | 2.66 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessed PTSD Checklist-5 (CAPS-5): Change in Mean Total Severity Scores From Baseline to 3-months Post-intervention
Description: Clinician-Administered PTSD Scale for DSM-5 also known as CAPS-5 is the gold standard in PTSD assessment. The CAPS-5 is a structured interview that was used to assess current (past month) PTSD symptom severity. The CAPS-5 total symptom severity score is the sum of 20 items, each scored 0-4, to yield a score with a possible range of 0-80. Higher scores mean worse outcome.
Time Frame: Baseline to 3-Months Post-Treatment (3-m PT): 3-m PT data were collected 11-13 weeks after the final session of TCTSY and CPT cohorts, which began in the same week. TCTSY (10 weeks) 3-m PT data collection occurred 2 weeks prior to CPT (12 weeks).
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 39 | 27
score on a scale | -11.41 (12.32) | -14.48 (12.01)

2. Primary Outcome: PTSD Symptom Checklist-5 (PCL-5): Change in Mean Total Score From Baseline to 3-month Post-intervention
Description: The PTSD Symptom-Checklist -Version 5 (PCL-5) is a 20-item, self-report instrument that assesses the presence and severity of DSM-V PTSD symptoms in the last month. It was summed for a total severity score ranging from 0-80, with higher scores representing greater symptom severity (worse outcomes). Within group changes in mean total PCL-5 score from baseline to 3-month post-intervention are reported here.
Time Frame: as for outcome 1
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 39 | 27
score on a scale | -9.99 (18.6) | -13.22 (17.39)

3. Secondary Outcome: Health-related Quality of Life: VR12, Mental Component Summary (MCS): Change in Mean MCS From Baseline to 3-month Post-intervention
Description: The VR-12 is a12-item self-rating scale that assess health-related quality of life in veterans and includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Results are expressed in terms of two meta-scores: the Mental Component Summary and the Physical Component Summary. The Mental Component Score (MCS) measures mental aspects of quality of life and ranges from 0 (extremely poor mental health) to 100 (extremely good mental health). The VR-12 is veteran population-normed with each component to have a mean score of 50 and a standard deviation of 10. Scores greater than 50 represent above average health status (better outcomes). The change in the mean MCS from baseline to 3-months post-treatment are presented here.
Time Frame: as for outcome 1
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 28
score on a scale | 4.92 (13.26) | 7.14 (9.15)

4. Secondary Outcome: Health-related Quality of Life: VR12, Physical Component: Change in Mean Subscale Score From Baseline to 3-month Post-intervention
Description: The VR-12 is a 12-item self-rating scale that assess health-related quality of life in veterans and includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Results are expressed in terms of two meta-scores: the Physical Component Summary and the Mental Component Summary. The Physical Component Score (PCS) measures physical aspects of quality of life and ranges from 0 (extremely poor physical health) to 100 (extremely good physical health), thus has a possible range of 0-100. The VR-12 is veteran population-normed with each component to have a mean score of 50 and a standard deviation of 10. Scores greater than 50 represent above average health status (better outcomes).
Time Frame: as for outcome 1
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 27
score on a scale | -2.74 (8.34) | -2.04 (9.68)

5. Secondary Outcome: BPI Pain Severity: Change in Total Severity Score From Baseline to 3-months Post-intervention
Description: The Brief Pain Inventory (BPI) contains three questions regarding pain severity. Pain severity is measured according to the worst pain experienced in the last three days, average pain in the last three days, and current pain; with each rated on an ordinal scale from "0" = "no pain" to "10" = "pain as bad as you can imagine." The pain severity score is the mean of the three pain severity item scores, with a potential range of 0-10; higher scores indicate worse outcomes.
Time Frame: as for outcome 1
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 34 | 23
score on a scale | 0.17 (1.66) | 0.30 (1.42)

6. Secondary Outcome: BPI Pain Interference: Change in Total Interference Score From Baseline to 3-months Post-intervention
Description: The Brief Pain Inventory (BPI) contains seven questions regarding pain interference that are rated on an ordinal numerical scale with anchors of 0 (no pain/interference) to 10 (maximum pain/interference). Pain interference assesses how that pain has affected general activity, mood, walking ability, normal work, relations with others, sleep, and enjoyment of life. The pain interference score is the mean of the seven pain interference item scores, with a potential range of 0-10; higher scores indicate worse outcomes.
Time Frame: as for outcome 1
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 34 | 23
score on a scale | 0.09 (2.41) | 0.12 (2.07)

7. Secondary Outcome: Changes in C-reactive Proteins (CRP) From Baseline to 3-months Post-intervention; Within Group Changes; Primary Site Only
Description: C-reactive protein (CRP) is a non-specific marker of inflammation. Blood samples of 25 ml were drawn into EDTA-containing (purple top) tubes and stored in a -80o freezer until analysis. The normal range is 8-10 mg/L. Higher levels of CRP indicate worse outcomes. The unit of analysis is the natural log (LN) of raw data (mg/L).
Time Frame: Baseline to 3-Months Post-Treatment (3-m PT): 3-m PT data were collected 11-13 weeks after the final session of TCTSY and CPT cohorts, which began in the same week.
Population: ITT sample with both baseline and 3-months post-intervention data. Some participants were lost to attrition. Sample is from primary site (Atlanta) only.
Measure: Mean (Standard Deviation); unit: LN(mg/L)
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 21 | 16
LN(mg/L) | -0.02 (0.76) | 0.17 (0.58)

8. Secondary Outcome: Changes in IL-6 Pro-inflammatory Cytokine From Baseline to 3-months Post-intervention; Primary Site Only
Description: IL-6 is a pro-inflammatory cytokine. Blood samples of 25 ml were drawn into EDTA-containing (purple top) tubes and stored in a -80o freezer until analysis. The normal range is < 5.0 pg/mL. Higher values indicate more inflammation (worse outcomes). The unit of analysis in these results is the natural log (LN) of the value (pg/mL).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: LN(pg/mL)
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 21 | 16
LN(pg/mL) | -0.30 (1.23) | 0.01 (1.12)

9. Secondary Outcome: Changes in IL-10 Anti-inflammatory Cytokine From Baseline to 3-months Post-intervention; Primary Site Only
Description: IL-10 is an anti-inflammatory cytokine. Blood samples of 25 ml were drawn into EDTA-containing (purple top) tubes and stored in a -80o freezer until analysis. The range of normal values is 4.8 - 9.8 pg/mL. Values out of range can indicate inflammatory dysregulation.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: LN(pg/mL)
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 21 | 16
LN(pg/mL) | 0.42 (1.75) | 0.18 (1.18)

10. Secondary Outcome: Changes in the Beck Depression Inventory-II (BDI-II) Total Score From Baseline to 3-months Post-intervention (Within Group)
Description: The Beck Depression Inventory II (BDI-II) is a 21-question multiple-choice self-report inventory widely used for assessing the severity of depression. The BDI-II total score is the sum of the 21 items, with a possible range of 0-63. Higher scores indicate worse outcomes.
Time Frame: as for outcome 7
Population: Some participants had missing or incomplete scale data, and some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 37 | 28
score on a scale | -6.89 (9.68) | -9.70 (10.37)

11. Secondary Outcome: Changes in the Difficulties in Emotion Regulation Scale (DERS) Total Score From Baseline to 3-months Post-intervention (Within Group)
Description: The Difficulties in Emotion Regulation Scale (DERS) is a brief, 36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation. The measure yields a total score as well as scores on six scales derived through factor analysis. The DERS total score is the mean of the 36 items score, with a potential range of 0-100. High scores indicate worse outcomes.
Time Frame: as for outcome 7
Population: Some participants had missing or incomplete scale data, and some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 39 | 25
score on a scale | -6.64 (24.95) | -15.68 (18.91)

12. Secondary Outcome: Changes in the PROMIS v2.0 Ability to Participate in Social Roles and Activities - Short Form 4a T-score From Baseline to 3-months Post-intervention (Within Group)
Description: Change in the PROMIS v2.0 - Ability to Participate in Social Roles and Activities -Short Form 4a (T-score) assesses the perceived ability to perform usual social roles and activities. Four items are worded negatively and are scored on a 5-point scale (5=never to 1= always). Responses are reverse-coded so that higher scores represent fewer limitations (better abilities). PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. Within group differences in T-scores (change scores) from baseline to 3-month follow up (3-month follow up T-score minus baseline T-score) were calculated. Positive change scores are indicative of improvement in perceived ability to participate in social roles and activity at the study endpoint.
Time Frame: as for outcome 7
Population: Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 28
T-score | 1.62 (6.92) | 3.29 (6.67)

13. Secondary Outcome: Changes in the PROMIS v2.0 Emotional Support 4a T-score From Baseline to 3-months Post-intervention (Within Group)
Description: The PROMIS v2.0 - Emotional Support 4a measure contains 4 items that assess perceived feelings of being cared for, valued, and having confidant relationships. Items are scored on a 5-point scale. Scores higher than 50 indicate more emotional support than the population mean. PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. Within group differences in T-scores (change scores) from baseline to 3-month follow up were calculated (3-month follow up T-score minus baseline T-score). Positive change scores are indicative of improvement in perceived emotional support at the study endpoint.
Time Frame: as for outcome 7
Population: Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 28
units on a scale | 0.60 (6.25) | 2.78 (7.64)

14. Secondary Outcome: Changes in the PROMIS v2.0 Satisfaction With Social Roles and Activities 4a T-score From Baseline to 3-months Post-intervention (Within Group)
Description: The 4-item PROMIS v2.0 - Satisfaction with Social Roles and Activities 4a was administered to participants at baseline and at 3-months post-intervention. The measure assesses satisfaction with performing social roles and activities. Items are scored on a 5-point scale and then reverse coded so that higher scores reflect great abilities to participate. Scores higher than 50 indicate higher perceived satisfaction than the population mean i.e., better outcomes. PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. Within group differences in T-scores (change scores) from baseline to 3-month post-intervention were calculated (3-month follow up T-score minus baseline T-score). Positive change scores are indicative of improvement in satisfaction with social roles and activities at the study endpoint.
Time Frame: as for outcome 7
Population: Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 28
units on a scale | 1.92 (6.82) | 2.55 (8.87)

15. Secondary Outcome: Changes in the PROMIS v2.0 Social Isolation 4a T-score From Baseline to 3-months Post-intervention (Within Group)
Description: The PROMIS v2.0 - Social Isolation 4a includes 4 items that assess feelings of isolation, companionship, and trust. The items scored on a five-point scale ("never" to "always"). PROMIS measure scores are computed to a T-score, where 50 represents the mean for US general population, and 10 is the standard deviation. Scores higher than 50 indicate more social isolation, i.e. worse outcomes. Within group differences in T-scores (change scores) from baseline to 3-month post-intervention were calculated (3-month follow up T-score minus baseline T-score). Positive change scores are indicative of increased social isolation at the study endpoint; negative change scores indicate decreased social isolation (better outcomes).
Time Frame: as for outcome 7
Population: Some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 40 | 28
units on a scale | -1.26 (7.80) | -2.65 (7.17)

16. Secondary Outcome: Changes in the Pittsburgh Sleep Quality Index Total Score From Baseline to 3-months Post-intervention (Within Group)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report scale consisting of 19 items that produce a global sleep quality score and the following 7 component scores: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction. Total score is reported here and has a potential range of 0-21. Higher scores indicate poorer sleep quality.
Time Frame: as for outcome 7
Population: Some participants had missing or incomplete scale data, and some participants were lost to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 37 | 28
score on a scale | -0.57 (3.30) | -2.32 (3.30)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at every data collection time point following baseline data collection, i.e. mid-intervention (weeks 5-6), 2-weeks post-intervention (weeks 12-14), and 3-months post-intervention (weeks 22-24). In addition, any adverse events that were spontaneously reported were documented.
Description: Anticipated adverse events are distinct from unanticipated adverse events for IRB purposes.
Arm/Group | Trauma Center Trauma-Sensitive Yoga (TCTSY) | Cognitive Processing Therapy (CPT)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/59
Other Adverse Events (participants affected / at risk) | 0/72 | 0/59

LIMITATIONS AND CAVEATS:
The study end point of three months post-treatment precluded determination of even longer-term sustained effects of the interventions. The CAPS-5 assessors were not blinded, introducing a risk of bias. The final cohort at Site 1 and the only cohort at Site 2 were conducted in 2020 during the COVID-19 pandemic, resulting in a pivot of study procedures to virtual delivery - which potentially confounded study data during that time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT02640690/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT02640690/ICF_001.pdf